CLINICAL TRIAL: NCT00975013
Title: Losing More Than Just Weight: Bone Loss After Laparoscopic Roux-en-Y Gastric Bypass
Brief Title: Bone Loss After Laparoscopic Roux-en-Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Principal Investigator, Kara Kallies, Academic Researcher, Gundersen Lutheran Medical Foundation
Other Study IDs: 2-07-02-009
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Bone Loss; Bone Density; Gastric Bypass; Bariatric Surgery
Keywords: Laparoscopic Gastric Bypass; Morbid Obesity; Bone Mineral Density
MeSH Terms: conditions — Bone Diseases, Metabolic; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

GROUPS / COHORTS (1):
- Bone Density Study Group: Morbidly obese, (BMI >40 kg/m2, or 35 kg/m2 with comorbidities) female patients who have given consent to undergo additional testing including bone densitometry, and lab testing preoperatively and at 6 and 12 months after undergoing elective laparoscopic roux-en-Y gastric bypass.

SUMMARY:
The objective of this study is to assess changes bone mineral density and bone metabolism after laparoscopic Roux-en-Y gastric bypass surgery. The investigators hypothesize that weight loss after laparoscopic Roux-en-Y gastric bypass surgery will be associated with increased bone turnover, changes in bone metabolism, and loss of bone mass.

DETAILED DESCRIPTION:
Obesity is an increasing problem within the United States. Fifteen million people in the United States are considered morbidly obese, with a body mass index (BMI) greater than 40 kg/m2. A wealth of literature has shown laparoscopic Roux-en Y gastric bypass surgery to be an effective procedure to reduce excess body weight. But a paucity of research examines the effects of laparoscopic Roux-en Y surgery on the skeleton.

Bone remodeling is a complex process involving bone resorption and formation-a process dependent upon local and systemic influences. Obesity is one of these influences that is poorly understood. Obesity is associated with a reduced risk of osteoporosis. Obesity may be protective due to increased weight bearing, increased production of estrogen by adipose tissue, or increased bone formation due to higher levels of insulin.

It is known that weight loss in healthy individuals is associated with bone loss. Several small studies have reported bone loss in patients undergoing vertical band gastroplasty or jejunoileal bypass weight loss surgeries. Other reported metabolic disease disarrangements following weight loss surgery are decreased serum calcium, decreased serum 25-hydroxy vitamin D, and hyperparathyroidism.

In the bariatric literature, weight loss has been associated with an increased risk of bone mineral loss and fracture. Osteoporosis has been described in patients who lost weight after jejunoileal bypass surgery. Premenopausal women appeared to be spared from bone mineral loss, thus indicating a protective effect from the premenopausal state. Bone mineral loss is seen both in premenopausal women and in men after weight loss surgery.

Roux-en Y gastric bypass has been shown to be more effective at weight loss than has the adjustable silicone gastric band. It has also been linked with increased loss of bone mineral density. Another study found an increase in bone turnover as well as a decrease in total bone mass and trochanteric bone density in laparoscopic Roux-en Y gastric bypass patients.

Previous research at our institution has shown a statistically significant increase in the prevalence of hyperparathyroidism in post-gastric bypass patients. However, our previous research did not examine the impact that these hormonal changes impart upon bone density. We have found a statistically significant incidence of vitamin D deficiency in our patients following this surgery. We intend to expand upon our own research as well as that of others by exploring the associations between the development of hyperparathyroidism, bone metabolic derangements, weight loss, and bone density.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese female patients undergoing elective laparoscopic Roux-en-Y gastric bypass at a single institution

Exclusion Criteria:

* Male patients
* Patients unable to fulfill the study protocol requirements

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of patients undergoing laparoscopic gastric bypass at a community-based teaching institution
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluate bone densitometry and lab tests to assess changes in bone mass and bone turnover after laparoscopic gastric bypass surgery | preoperatively and at 6 and 12 months after laparoscopic Roux-en-Y gastric bypass

SECONDARY OUTCOMES:
Evaluate weight loss, menopausal and nutritional status to assess correlations with results from bone densitometry and lab values after laparoscopic gastric bypass surgery | preoperatively, and at 6 and 12 months after laparoscopic Roux-en-Y gastric bypass

CONTACTS AND LOCATIONS:
Overall Officials: Shanu N Kothari, M.D., Principal Investigator — Gundersen Lutheran Health System; Kevin P Riess, M.D., Principal Investigator — Gundersen Lutheran Medical Foundation; Current Practice: SMDC Health System-Duluth Clinic
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] Morberg CM, Tetens I, Black E, Toubro S, Soerensen TI, Pedersen O, Astrup A. Leptin and bone mineral density: a cross-sectional study in obese and nonobese men. J Clin Endocrinol Metab. 2003 Dec;88(12):5795-800. doi: 10.1210/jc.2003-030496. PMID 14671171
- [Background] Cundy T, Evans MC, Kay RG, Dowman M, Wattie D, Reid IR. Effects of vertical-banded gastroplasty on bone and mineral metabolism in obese patients. Br J Surg. 1996 Oct;83(10):1468-72. doi: 10.1002/bjs.1800831046. PMID 8944476
- [Background] von Mach MA, Stoeckli R, Bilz S, Kraenzlin M, Langer I, Keller U. Changes in bone mineral content after surgical treatment of morbid obesity. Metabolism. 2004 Jul;53(7):918-21. doi: 10.1016/j.metabol.2004.01.015. PMID 15254887
- [Background] Meyer HE, Tverdal A, Selmer R. Weight variability, weight change and the incidence of hip fracture: a prospective study of 39,000 middle-aged Norwegians. Osteoporos Int. 1998;8(4):373-8. doi: 10.1007/s001980050077. PMID 10024908
- [Background] Bano G, Rodin DA, Pazianas M, Nussey SS. Reduced bone mineral density after surgical treatment for obesity. Int J Obes Relat Metab Disord. 1999 Apr;23(4):361-5. doi: 10.1038/sj.ijo.0800827. PMID 10340813
- [Background] Coates PS, Fernstrom JD, Fernstrom MH, Schauer PR, Greenspan SL. Gastric bypass surgery for morbid obesity leads to an increase in bone turnover and a decrease in bone mass. J Clin Endocrinol Metab. 2004 Mar;89(3):1061-5. doi: 10.1210/jc.2003-031756. PMID 15001587
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Background] Carlin AM, Rao DS, Yager KM, Parikh NJ, Kapke A. Treatment of vitamin D depletion after Roux-en-Y gastric bypass: a randomized prospective clinical trial. Surg Obes Relat Dis. 2009 Jul-Aug;5(4):444-9. doi: 10.1016/j.soard.2008.08.004. Epub 2008 Aug 14. PMID 18996761